CLINICAL TRIAL: NCT06467110
Title: A Prospective, Multicenter, Single-Arm Clinical Trial to Assess the Safety and Efficacy of a Transcatheter Mitral Valve Clip Delivery System With Steerable Guide Catheter in Patients With Moderate-Severe or Severe Degenerative Mitral Regurgitation (DMR)
Brief Title: Safety and Effectiveness Study of SQ-Kyrin TMVr System for Degenerated Mitral Regurgitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVRP01-001B
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2023-07

CONDITIONS: Degenerated Mitral Regurgitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transcatheter mitral valve clip delivery system and steerable guide catheter (Shenqi Medical) (Experimental): The principle of this product is the transcatheter interventional edge-to-edge repair technology (edge-to-edge repair). The core technology is to treat the regurgitation by edge-to-edge suturing the mitral valve. The double holes are set in the mitral valve (A2/P2 zone) or the edges in A1/P1 or A3/P3 zones are apposed and closed to treat regurgitation.
  Interventions: Device: transcatheter mitral valve clip delivery system and steerable guide catheter (Shenqi Medical)

INTERVENTIONS:
Device: transcatheter mitral valve clip delivery system and steerable guide catheter (Shenqi Medical) — The principle of this product is the transcatheter interventional edge-to-edge repair technology (edge-to-edge repair). The core technology is to treat the regurgitation by edge-to-edge suturing the mitral valve. The double holes are set in the mitral valve (A2/P2 zone) or the edges in A1/P1 or A3/P3 zones are apposed and closed to treat regurgitation.

SUMMARY:
To verify the safety and effectiveness of transcatheter mitral valve clip delivery system and steerable guide catheter produced by Shanghai Shenqi Medical Technology Co., Ltd.in patients with moderate-severe or severe degenerated mitral regurgitation (DMR).

DETAILED DESCRIPTION:
This study is clinical research using a prospective, multicenter, single arm method to evaluate the safety and effectiveness of transcatheter mitral valve clip delivery system and steerable guide catheter transcatheter mitral valve clip delivery system and steerable guide catheter in the treatment of patients with moderate-severe (3+) or severe (4+) degenerated mitral regurgitation. A total of 118 subjects are planned to be included in this trial. All subjects are treated with transcatheter mitral valve clip delivery system and steerable guide catheter transcatheter mitral valve clip delivery system and steerable guide catheter, and are followed up at 30 days, 6 months and 12 months after surgery. At the follow-up of 12 months after surgery, the composite endpoints of no death, no surgical mitral valve related surgery due to mitral valve dysfunction, and no moderate-severe or severe MR (MR > 2 +) are evaluated. After the follow-up of 12 months after surgery, the stage statistical analysis, clinical summary and application for product registration are performed.

ELIGIBILITY:
Inclusion Criteria:

* Severe MR ≥3+ as determined by transthoracic echocardiography (TTE);
* STS risk score results show that patients at high risk for traditional surgery or patients who cannot tolerate traditional thoracotomy: Subjects judged to be refractory to mitral valve surgery due to a ≥ 8% risk of death from STS surgery for surgical mitral valve replacement, or a ≥ 6% risk of death from STS surgery for surgical mitral valve repair, or because of any of the following risk factors:

  1. Porcelain aorta or active ascending aortic plaque
  2. Mediastinum treated with radiotherapy
  3. Past mediastinitis
  4. Left ventricular ejection fraction (LVEF) <40%
  5. Presence of a patent coronary bypass implant
  6. Acceptance of two or more cardiothoracic surgeries
  7. Liver cirrhosis
  8. Other surgical risk factors
* Patients with Degenerated MR (Degenerated MR);
* Age ≥ 18 years old, regardless of gender;
* Classification of cardiac function: NYHA class II, III or ambulatory class IV;
* Patients assessed by a multidisciplinary cardiac team as very high-risk or unsuitable for routine mitral valve surgery;
* Be able to understand the objective of the trial, and volunteered to participate and signed the Informed Consent Form, willing to accept the relevant examination and clinical follow-up.
* Left ventricular end-systolic diameter (LVESD)≤60mm
* The MR beam mainly originates from the A2/P2 area
* Mitral valve disease prolapse lesion area width≤15mm, prolapse height≤10mm, effective length of anterior and posterior valve leaflets>10mm
* Mitral valve effective orifice area (EOA) ≥ 4.0cm2
* No obvious calcification of mitral valve leaflets
* Patient anatomy allows atrial septum approach

Exclusion Criteria:

* History of mitral valve surgery;
* Patients with infective endocarditis or suggestive of active infection;
* Complicated with severe untreated coronary artery disease;
* Patients with pulmonary hypertension (pulmonary systolic blood pressure>70mmHg);
* Patients with transthoracic echocardiographic evidence suggesting moderate-severe to severe right ventricular dysfunction;
* Left ventricular ejection fraction <20%;
* Patients who are extremely frail and cannot tolerate general anesthesia surgery or is in the state of shock requiring circulatory support;
* Patients diagnosed with hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis;
* Mitral regurgitation due to active rheumatic heart disease or rheumatic etiology;
* Severe renal insufficiency (eGFR ≤ 25 mL/min) or requiring chronic renal replacement therapy;
* Patients with definite coagulation disorders and severe coagulation system diseases;
* Patients with clear contraindications to the use of anticoagulants;
* Patients with stroke or transient cerebral ischemic attack within 30 days;
* Any intracardiac mass, left ventricular or atrial thrombus detected on transthoracic echocardiography;
* Severe tricuspid TR;
* Patients with other valve disease requiring surgery or interventional therapy;
* Patients with severe macrovascular disease requiring surgical treatment;
* Severe symptomatic carotid stenosis (>70% on ultrasonography) or carotid stenting within 30 days;
* Patients with inappropriate anatomical structures of the heart and valves indicated by imaging examinations;
* Known allergy to contrast agents and nickel-titanium memory alloy products;
* R<testing systolic blood pressure 90 mmHg or >160 mmHg;
* Patients with diseases that seriously affect the evaluation of treatment, such as patients with severe neurological lesions affecting cognitive ability, patients with malignant tumors, etc.;
* Patient life expectancy < 12 months;
* Patients with severe thoracic deformity;
* Women who are pregnant, breastfeeding, or planning to become pregnant within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of composite endpoint of no death, no surgical mitral valve-related procedures due to mitral valve dysfunction, and no moderate-severe or severe MR (MR>2+) at 12 months after surgery | 12 months after surgery
  Incidence of composite endpoint of no death, no surgical mitral valve-related procedures due to mitral valve dysfunction, and no moderate-severe or severe MR (MR>2+) at 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, PLA, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No